CLINICAL TRIAL: NCT03863522
Title: Automated Method for Breast Cancer Detection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate FNA samples (low cell counts)
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: J18138; IRB00172441 (Other: JHMI IRB)
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Breast Cancer Diagnosis
Keywords: Breast Cancer Diagnosis; Ultrasound-guided core needle biopsy; Fine needle aspiration; FNA; Diagnostic Cartridge
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fine Needle Aspiration (Other): Participants will receive fine needle aspiration (FNA) later read by the cytopathologist and the cartridge. All patients will receive standard of care (Ultrasound-guided core needle biopsy and diagnosis).
  Interventions: Procedure: Fine needle aspiration; Device: Cancer Detection cartridge

INTERVENTIONS:
Procedure: Fine needle aspiration — Fine needle aspiration is a type of biopsy procedure to diagnose suspicious lesions. After giving numbing medicine, a thin needle is inserted into the breast to obtain a sample. This procedure is followed by the standard of care and will last about 10 minutes. The sample will be analyzed by a diagnostic cartridge and by the cytopathologist.
  Other Names: FNA
Device: Cancer Detection cartridge — The Cancer Detection cartridge has the ability to measure methylated gene changes in breast cells. The device will not be in contact with the patients. The FNA samples will be smeared on a slide which will be placed into the cartridge for analysis.

SUMMARY:
Participants with suspicious breast lesions by mammography will undergo fine needle aspiration (FNA) under ultrasound guidance. The FNA will be read by the cytopathologist and analyzed in the breast cancer detection cartridge. All patients will receive standard of care (Ultrasound-guided core needle biopsy and diagnosis). We will also receive FNA collected from 60 patients with palpable lesions in South Africa and analyze them samples in our lab with the same method.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be female
* Patient must be 18 years of age or older
* Patient has been recommended for ultrasound core needle biopsy of a suspicious breast lesion

Exclusion Criteria:

* Patients may be excluded for any condition that in the opinion of the investigator may not make it safe to take part (e.g. certain medicines).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2019-03-07 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Mullen, MD, Principal Investigator — JHU School of Medicine
Locations (2):
- United States (2):
  - Johns Hopkins Hospital Outpatient Center, Baltimore, Maryland
  - Johns Hopkins Medical Imaging at Green spring Station, Lutherville-Timonium, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fine Needle Aspiration
Started | 116
Completed | 116
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 116
Age, Continuous [Mean (Full Range); unit: years] | 48 [18 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 71
  White | 40
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 62
  South Africa | 54

OUTCOME MEASURES:

1. Primary Outcome: Correlation of Diagnostic Cartridge With Histopathology as Assessed by Number of Participants With Same Diagnosis From Both Cancer Detection Cartridge and Core Biopsy or Resected Lesion
Description: Number of participants in whom DNA methylation profile of 10 genes in the Cancer Detection cartridge correlates with diagnosis based on the gold standard of histopathology of the core biopsy or resected sample.
Time Frame: up to 2 years
Population: Inadequate cell counts prevented analysis of samples. Data was not generated.
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 0

2. Primary Outcome: Correlation of Diagnostic Cartridge With Cytopathology as Assessed by Number of Participants With Same Diagnosis From Both Cancer Detection Cartridge and Cytology of Fine Needle Aspiration (FNA)
Description: Number of participants in whom DNA methylation profile of 10 genes as determined in the Cancer Detection cartridge correlates with FNA cytology
Time Frame: up to 2 years
Population: Inadequate cell counts prevented analysis of samples. Data was not generated.
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 0

3. Secondary Outcome: Correlation of Diagnostic Cartridge With Known Lab Assay
Description: Number of participants in whom gene-methylation prediction of FNA in the Cancer Detection cartridge is malignant or benign when compared to gene-methylation prediction of FNA using our known laboratory assay (QM-MSP)
Time Frame: up to 2 years
Population: Inadequate cell counts prevented analysis of samples. Data was not generated.
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 0

4. Secondary Outcome: Correlation of Known Lab Assay for FNA Versus the Core Biopsy
Description: Number of participants in whom gene-methylation prediction of benign or malignant using our known laboratory assay (QM-MSP) matches for both the FNA sample and the core biopsy sample
Time Frame: up to 2 years
Population: Inadequate cell counts prevented analysis of samples. Data was not generated.
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 0

5. Secondary Outcome: Correlation of Cartridge Based Quantitative Evaluation of Tumor Markers (ER/PR/Her2 and Ki67) in FNA Versus FFPE Sections
Description: Number of participants with same expression of ER/PR/Her2 and Ki67 in FNAs of methylation positive breast lesions as with expression of ER/PR/Her2 and Ki67 in Formalin-Fixed Paraffin-Embedded (FFPE) sections of tumors using cartridge based quantitative evaluation
Time Frame: up to 2 years
Population: Inadequate cell counts prevented analysis of samples. Data was not generated.
Arm/Group | Fine Needle Aspiration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The only intervention is FNA, which is immediately preceded by a core needle biopsy. Thus the cause, FNA vs core biopsy, of the AE will be impossible to determine. Via phone 1-2 days post-procedure and again 10-14 days post-procedure, patients were asked about any bruising and pain, but could report other symptoms if any. Please note only the 62 Johns Hopkins patients were called; the remaining 54 South African patients were not followed for AEs by this study team.
Arm/Group | Fine Needle Aspiration
All-Cause Mortality (participants affected / at risk) | 0/62
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 3/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fine Needle Aspiration (N=62)
Bruising (Injury, poisoning and procedural complications) | 0 (0)
Pain (Injury, poisoning and procedural complications) | 3 (3)
Other (Injury, poisoning and procedural complications) | 0 (0) — Any other self-reported symptom

LIMITATIONS AND CAVEATS:
Enrollment was halted early due to the quality of samples obtained. Samples contained insufficient cells and could not be analysed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03863522/Prot_SAP_001.pdf